CLINICAL TRIAL: NCT05043181
Title: Exosome-based Nanoplatform for Ldlr mRNA Delivery in Familial Hypercholesterolemia
Brief Title: Exosome-based Nanoplatform for Ldlr mRNA Delivery in FH
Acronym: ENDFH
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Lijun Yuan, MD, PhD, Director of the department of ultrasound diagnostics, Tang-Du Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210817V2.0
Record Dates: First submitted 2021-09-03; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Homozygous Familial Hypercholesterolemia (Experimental)
  Interventions: Biological: Low Density Lipoprotein Receptor mRNA Exosomes

INTERVENTIONS:
Biological: Low Density Lipoprotein Receptor mRNA Exosomes — The study consists of two phases: dose escalation phase and extension phase. Dose escalation phase：For the intervention of low-density lipoprotein receptor mRNA (LDLR mRNA) exosomes. A total of six dose groups are planned, with single dose of 0.044 mg/kg, 0.088 mg/kg, 0.145 mg/kg, 0.220 mg/kg, 0.295 mg/kg and 0.394 mg/kg, respectively. About 3 subjects are enrolled in each dose group. In the 0.044 mg/kg group, the second and third subjects are required to start exosome infusion treatment after the treatment of the previous subjects, and the other dose groups are not required to do this. There are three treatments in total, and the interval between each exosome treatment is 7±1 d.
  Extension phase: About 12 subjects are further enrolled. The subjects will receive 3 intravenous/peritoneal infusion treatment of LDLR mRNA exosomes once a week for three weeks, whose single dose is determined in the dose escalation phase.

SUMMARY:
mRNA therapy is a highly promising gene therapeutic strategy in the treatment of Homozygous Familial Hypercholesterolemia (HoFH). Exosomes is safe and efficient carriers for mRNA drug delivery, due to their biocompatibility, bioavailability. This first-in-human study is aimed to evaluate the safety and preliminary effectiveness of Exosome-based ldlr mRNA nanoplatform for gene therapy in HoFH.

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is an autosomal dominant genetic disease characterized by severely elevated plasma low-density lipoprotein (LDL) cholesterol (LDL-C) and premature coronary heart disease. Most of FH patients (about 95% of cases) are attributed to functional loss mutation of the LDL receptor (LDLR) gene. The prevalence of the heterozygous mutations in LDLR has been estimated at 1 in 200 to 1 in 500 in the population, and the homozygous form in 1 in 100000 individuals. As a key lipoprotein receptor on the surface of hepatocyte, the LDLR is critical for liver clearing LDL-C from the circulation. By endocytosis and further processing of the LDL-C, LDLR is responsible for removing most excess LDL-C from the serum, and there are no substitutes in vivo. These heterozygotes (HeFH) typically have twice the normal plasma LDL levels and cardiovascular diseases at an earlier age. Homozygous individuals (HoFH) face much higher LDL-C levels and often die before the age of 20 years if untreated. Although existing therapeutics, such as statins, ezetimibe and PCSK9 inhibitors, have some beneficial effects on HeFH, few drugs have therapeutic effects on HoFH even at high-doses. Lipid apheresis and liver transplantation are the current clinical managements to reduce the LDL-C level, while gene therapy holds the promise.

Exosomes are small intracellular vesicles ranging in 30-150 nm size and have an important role in cell-cell communication. Many studies show that exosome can efficiently deliver cargos, such as mRNA, miRNA and even plasmid DNA, to target cells, emerging as a promising therapeutic carrier for gene therapy. Compared with virus, exosomes, as "natural nanoparticles", are easy to handle, non-cytotoxic and non-immunogenic. It is thus promising to develop exosome-based LDLR-gene delivery strategy and explore the therapeutic effects on HoFH.

In this study, an Ldlr-expressing virus vector will be constructed to generate Ldlr mRNA-enriched exosomes. To meet the standards of clinical trials, we will use the GMP-grade compliant normal donor bone marrow-derived MSCs to produce exosomes. Exosomes will be enriched by filtration and ultracentrifugation, and then normalized by Nanosight, Electron microscopy and key exosomes biomarkers. In order to ensure the safety of patients, we plan to inject exosomes through abdominal puncture under ultrasound guidance, and purchase medical insurance for patients. This first-in-human study is aimed to evaluate the safety of this exosome product for gene therapy and preliminary evidence of efficacy using plasma LDL-C levels as a surrogate biomarker. The study is promising to provide a new therapeutic approach for the treatment of Homozygous Familial Hypercholesterolemia patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45, no gender limitation;
2. Patients with homozygous familial hypercholesterolemia diagnosed by genetic testing.
3. Understand the study and be willing to participate in the study with the informed consent signed

Exclusion Criteria:

1. those who have severe comorbidities, including any of the following: A) unstable angina pectoris and/or congestive heart failure requiring hospitalization; B) myocardial infarction or cerebrovascular accident within the last 6 months; C) chronic obstructive pulmonary disease worsens or requires hospitalization; D) serious diseases of vascular, nervous system, blood, gastrointestinal and endocrine systems or metabolic disorders; E) autoimmune/immune deficiency diseases such as rheumatoid arthritis, acquired immune deficiency syndrome, and so on; F) malignant tumor or other chronic infection.
2. those who previously received targeted drug therapy, cell therapy, gene therapy or others immunotherapy;
3. those who had organ transplants in the past;
4. any of the following abnormalities are found in the laboratory examination: A) blood routine examination: absolute neutrophil count (ANC) < 1.5×109/L, or platelet (PLT) < 50×109/L, or hemoglobin (HGB) < 80 g/dL; B) coagulation function: prothrombin time (PT), or activated partial thrombin time (APTT), or INR > 1.5×ULN; C) liver function: total bilirubin (TBIL) > 2×ULN (upper limit of normal value), or alanine transferase (ALT), aspartate transferase (AST), alkaline phosphatase (ALP) > 5×ULN; D) renal function: serum creatinine (Cr) ≥1.5×ULN, or glomerular filtration rate (GFR) < 60 mL/min·1.73m2; E) cardiac ultrasound: left ventricular ejection fraction (LVEF) < 50%.
5. those who are known or expected to have an allergic reaction to or have a history of allergic reaction to any of the ingredients treated by this test;
6. those who have a history of contrast agent allergic;
7. those who have a clear history of mental disorders in the past;
8. those who have a history of drug abuse or drug use;
9. Pregnant or lactating women;
10. Women of childbearing age and fertile men cannot take effective and adequate contraceptive measures (such as intrauterine device (IUD), condom, spermicidal gel plus condom, uterine cap, etc.) during the period of receiving the study drug and 3 months after the end of the study;
11. those who participated in the clinical study of other drugs within 3 months before joining the group;
12. Subjects that are not suitable to participate in this study for other reasons judged by the investigators.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes of Total Cholesterol | Changes from Baseline Total Cholesterol at Day 19
  mmol/L
Changes of Low-Density Lipoprotein Cholesterol | Changes from Baseline Low-Density Lipoprotein Cholesterol at Day 19
  mmol/L
Changes of High-Density Lipoprotein Cholesterol | Changes from Baseline High-Density Lipoprotein Cholesterol at Day 19
  mmol/L
Changes of Triglyceride | Changes from Baseline Triglyceride at Day 19
  mmol/L

SECONDARY OUTCOMES:
Changes of Degree of Coronary Stenosis | Changes from Baseline Degree of Coronary Stenosis at Day 28
  % determined by coronary CT
Changes of Volume of Carotid Artery Plaques | Changes from Baseline Volume of Carotid Artery Plaques at Day 28
  cm3 determined by ultrasound
Changes of Stability of Carotid Artery Plaques | Changes from Baseline Stability of Carotid Artery Plaques at Day 28
  Grade I, II, III determined by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Lijun Yuan, Principal Investigator — Tangdu Hospital-Air Force Medical University
Locations (1):
- Tangdu Hospital, Air Force Medical University, Xi'an, Shannxi, China